CLINICAL TRIAL: NCT06584513
Title: Implementing a Patient-centred and Evidence-based Intervention to Reduce BEnzodiazepine and Sedative-hypnotic Use to Improve Patient SAFEty and Quality of Care (BE-SAFE)
Brief Title: Improving Patient Safety by Supporting Older Adults in Managing Sleep Problems.
Acronym: BE-SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Oslo University Hospital (Other); National and Kapodistrian University of Athens (Other); Institute of Psychiatry and Neurology, Warsaw (Other); CHU UCL Namur (Unknown); Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-00702
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Benzodiazepines Deprescribing; Sleep Problems
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Participating physicians will be randomly assigned in a 1:1 ratio in clusters to either the intervention group or the control group. Patients of participating physicians will be assigned to the physician randomisation group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessment is performed by research team blinded to the allocated intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician and patient intervention (Experimental): Patients in the intervention group will be treated by physicians, who received informative and educative materials (including videos) and training, including guidelines and implementation recommendations on how to deprescribe, on shared-decision making with patients, on how to manage sleep problems using alternative methods other than BSH. Patients receive brochures and access to videos. Communication forms are implemented to ensure continuity of care.
  Interventions: Other: Specific tapering plan for sleep medication, educational and cognitive behavioural therapy elements
- Control/Usual care (No Intervention): Participants in the control group receive treatment according to standard care of the prescribing physician, who did not receive any training or additional material.

INTERVENTIONS:
Other: Specific tapering plan for sleep medication, educational and cognitive behavioural therapy elements — The intervention consists of a patient-centred intervention to help patients in deprescribing BSHs and better managing their sleep problems. The material used consists of training modules, brochures, and self-monitoring tools. There are materials for physicians and for patients.
  Arms: Physician and patient intervention

SUMMARY:
Among older adults (≥65 years), use of sleeping pills, such as benzodiazepines and other sedative-hypnotics, to treat sleep problems is common. While sleeping pills are effective in the first few weeks of use, their effect diminishes significantly after that. Especially older adults are susceptible to significant adverse effects of sleep pills, yet stopping sleeping pills remains challenging. BE-SAFE aims to conduct a randomised study testing a patient-centred intervention to reduce sleeping pill use and to improve patient safety and quality of care focusing on implementation aspects. The intervention addresses knowledge and practice gaps related to discontinuation of sleeping pills in older adults with sleep problems.

DETAILED DESCRIPTION:
Background:

Use of Benzodiazepine and Sedative Hypnotics (BSHs) is one of the three overuse practices measured by the OECD. BSH use has been reported to be as high as 15-30% in older adults with 87% taking BSHs for sleep problems. Use of BSHs is associated with significant adverse effects such as falls, fractures, hospitalisations, impaired functioning, delirium, dementia and mortality and therefore threatens patient safety. This applies especially to older adults as they are more susceptible to adverse effects due to changes in pharmacokinetics and pharmacodynamics associated with age and to the frequent presence of polypharmacy and comorbidities.

Design:

Multicenter, superiority (first co-primary endpoint) and non-inferiority (second co-primary endpoint) cluster randomised controlled trial (RCT) conducted in six countries across Europe (Belgium, Greece Norway, Poland, Spain, and Switzerland). Participating physicians will be randomly assigned in a 1:1 ratio in clusters to either the intervention group (with training and additional material to overcome sleeping problems and to help participants discontinue BSH) or the control group (treatment according to standard of care without training or additional material). Eligible patients will be enrolled with their treating physician defined as the cluster. Outcome assessment will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* BSH (ATC codes N05BA, N05CF, N05CD, and N03AE01) use on average ≥3 times a week during the last 3 months prior to providing informed consent, as self-reported by the patient or by the informal carer
* Taking BSH for sleep problems, as self-reported by the patient or by the informal carer

Exclusion Criteria:

* Indication for BSH appropriate or withdrawal dangerous, based on available documents (diagnosis list) or General Practitioner (GP) information:

  * Current use of BSH for alcohol withdrawal
  * BSH use in the context of addiction
  * Rapid Eye Movement (REM) sleep Behaviour Disorders
  * Active diagnosis of severe non-REM-related parasomnias with risk of self-damage or giving harm to others or with high frequency or social embarrassment
  * Epilepsy (all forms, because of risk of seizures by sleep deprivation)
  * Current active diagnosis of severe general or specific anxiety disorder (including obsessive compulsive disorder, social phobia, post-traumatic stress disorder, panic disorder with or without agoraphobia)
  * Current active diagnosis of psychotic disorder with or without antipsychotic medication
  * Current active diagnosis of severe depression with or without major anxiety symptoms
  * Current active diagnosis of bipolar disorder with or without major anxiety symptoms
  * Acute suicidal ideation
* Current formal active tapering process of BSHs supported by a physician
* Planned admission to palliative care within 24 hours of inclusion or estimated life-expectancy of less than 12 months i.e., patient is in a state or has a diagnosis where the cluster physician would not be surprised if patient dies within the next months (this criterion is relatively vague and subjective but because there is no validated prognostic score, it is justified)
* Inability to provide informed consent (e.g., because of cognitive impairment), except if a proxy can provide consent, be actively involved in the study, and patient shows no sign of disagreement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
BSH discontinuation | 12 months after enrollment
  Number of patients with BSH discontinuation according to self-/informal carer-disclosure. Discontinuation is defined as the intake of a maximum of one tablet within the previous 14 days.
Quality of sleep | 12 months after enrollment
  Quality of sleep measured by the Insomnia Severity Index (ISI). The questionnaire consists of 7 questions, answers range from 0-4 points, which are added up to get a total score. The higher the total score, the more severe level of insomnia.

SECONDARY OUTCOMES:
Use of a substitute medication for sleep | 2 months, 6 months, and 12 months after enrollment
  Use of a substitute medication for sleep, according to self-/informal carer disclosure
BSH discontinuation discussion with HCP | 1 month, 2 months, and 6 months after enrollment
  Number of patients who discussed BSH discontinuation with a HCP during the last month at M01 and M02, and during the last 4 months at M06
Benzodiazepines (BSH) discontinuation or dose reduction | 2 months and 6 months after enrollment
  Number of patients with BSH discontinuation or dose reduction, according to self-/informal carer disclosure. Defined as the intake of a maximum of one tablet within the previous 14 days.
BSH adverse events | 12 months after enrollment
  Number of patients with adverse effects of BSHs within 12 months of follow-up, according to self/informal carer disclosure, that is:
  * Falls leading to emergency room visit or hospitalisation
  * Fall-related fractures leading to emergency room visit or hospitalisation. As a sensitivity analysis, facial, fingers/toes, and ankle fractures that are less likely to be osteoporotic fractures will be excluded.
  * Delirium leading to emergency room visit or hospitalisation
  * Hospitalisations
  * Death from any cause
Quality of sleep | 2 months and 6 months after enrollment
  Quality of sleep measured by the Insomnia Severity Index (ISI). The questionnaire consists of 7 questions, answers range from 0-4 points, which are added up to get a total score. The higher the total score, the more severe level of insomnia.
BSH standardized daily dose intake | 2 months, 6 months, and 12 months after enrollment
  Standardized daily dose intake based on equivalent doses for BSH (lorazepam-equivalent).
Health-related quality of life | 2 months, 6 months, and 12 months after enrollment
  Health-related quality of life measured by the European Quality of Life-5 Dimensions questionnaire (EQ-5D-5L). Consists of a visual analogue scale and short descriptive system questionnaire, corresponding to 5 severity levels of health state, higher level indicating more severe problems.
Withdrawal symptoms from BSH discontinuation | 2 months and 6 months after enrollment
  Number of patients with withdrawal symptoms from BSH discontinuation measured by the Clinical Institute Withdrawal Assessment Scale (CIWA-B). Questionnaires composed of 20 questions, with scale that range from 0-4, which are added up to give a total score. Higher scores indicate more severe levels of withdrawal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD, MAS, Study Chair — University Hospital Bern (Inselspital)
Locations (6):
- Centre Hospitalier Universitaire CHU UCL Namur, Yvoir, Belgium
- National and Kapodistrian University of Athens, Athens, Greece
- Oslo University Hospital, Nydalen, Norway
- Institute of Psychiatry and Neurology, Warsaw, Poland
- Universitat Autònoma de Barcelona, Barcelona, Spain
- Department of General Internal Medicine, University Hospital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No